CLINICAL TRIAL: NCT06196502
Title: Effect of Gentle Human Touch and Kangaroo Care Applied During Hepatitis-B Vaccination in Newborns on Pain, Crying Duration and Physiological Parameters: Randomized Controlled Study
Brief Title: The Effect of Gentle Human Touch and Kangaroo Care on Pain and Crying Physiological Parameters During Hepatitis-B Vaccination in a Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Elif Tuba KOC, Child Health and Diseases Nursing Department President, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AhiEvranU-UTubaKOÇ-001
Record Dates: First submitted 2023-11-16; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: newborn; pain; intervention; pediatric nursing; vaccination
MeSH Terms: conditions — Pain | interventions — Kangaroo-Mother Care Method; Lactation

STUDY DESIGN:
Intervention Model Description: There are three sections to it, and they will all be finished simultaneously. This is not a study of drugs or devices. The three arms of the study are the breastfeeding (standard care), kangaroo care, and gentle human touch groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gentle human touch (GHT) (Experimental): Experimental: Gentle human touch (GHT) Group 1: Gentle touch is a touch technique that provides a kind of relaxation in premature babies, reduces behavioral stress and motor activities of babies and is effective in their positive behavior.
  Interventions: Other: Gentle Human Touch (GHT)
- Kangaroo Care (Active Comparator): Experimental: Kangaroo Care Group 2: Kangaroo care is a comforting technique that strengthens and bonds the baby and parent, increases the production of milk by the mother, and lessens the stress and anxiety of both parties. Kangaroo care between parent and baby is a method that regulates vital values, reduces the possibility of hypoglycemia and prevents hypothermia.
  Interventions: Other: Kangaroo Care
- Lactation (Active Comparator): Breastfeeding will begin 5 minutes before the Hepatitis-B vaccine administration and will continue during and after the procedure. It is planned to last 10 minutes in total.
  Interventions: Other: Lactation

INTERVENTIONS:
Other: Gentle Human Touch (GHT) — Gentle touch is a touch technique that provides a kind of relaxation in premature babies, reduces behavioral stress and motor activities of babies and is effective in their positive behavior. GHT Hepatitis-B vaccine will start 5 minutes before the application and continue during and after the procedure. It is planned to take 10 minutes in total. The researcher will place one hand on the baby's head and the other hand on the baby's lower abdomen, covering the waist and hips, for 10 minutes.
  Arms: Gentle human touch (GHT)
Other: Kangaroo Care — Kangaroo care will be provided to randomly selected volunteer moms in their own gynecological ward rooms, where they will have skin-to-skin contact with their babies while maintaining their privacy. Kangaroo care is a strategy that promotes bonding and engagement between a mother and her infant by allowing skin-to-skin contact with the newborn's face facing the mother and only the diaper remaining.
  The infant is positioned such that his or her shoulders are totally on the mother's chest, ensuring the baby's airway is open. To avoid heat loss while the baby is in skin-to-skin contact with his mother, a tiny blanket will be placed on his back and a beanie will be placed on his head. Kangaroo care will begin 5 minutes before the Hepatitis-B vaccine is administered and will continue throughout the operation. It is estimated that it will take 10 minutes in total.
  Arms: Kangaroo Care
Other: Lactation — Breastfeeding will become standard medical practice. Breastfeeding will start as soon as the baby is given the vaccination and continue throughout the process.
  Arms: Lactation

SUMMARY:
Many short- and long-term consequences, including altered physiological parameters, issues with feeding and sleep, chronic pain syndrome, difficulty focusing, anxiety, cognitive behavioral disorders, adjustment disorders, and growth retardation, have been linked to pain in neonates. Each and every newborn is entitled to pain relief and reduction. Avoiding painful interventions is the most crucial tactic in the management of newborn pain. However, it is impossible to ignore the necessity of therapeutic and diagnostic interventions. As such, pain reduction and elimination are crucial. Non-pharmacological techniques used on infants undergoing invasive operations have been shown in studies to be successful in reducing discomfort, pain, and restlessness while also enhancing comfort.

Numerous non-invasive, non-pharmacological techniques are employed for this goal. Among the non-invasive, non-pharmacological techniques include breastfeeding, nursing, therapeutic touch, skin-to-skin contact, wrapping, swaddling, music therapy, and white noise. The Hepatitis-B vaccine is among the first invasive therapies administered to infants. Research indicates that pain scores are positively impacted by canopy touch. Skin-to-skin contact is achieved by a number of techniques. The most popular is kangaroo care, which is given to mothers nude on their chests. Gentle human touch is another technique used to lessen pain during invasive operations (GHT). GHT is a soothing tactile stimulation that doesn't involve touching or rubbing. Several research have examined GHT's impact and discovered that it effectively reduces pain.

The purpose of this study was to ascertain how GHT and Kangaroo care affected the newborn's pain, length of crying, and physiological parameters while the Hepatitis-B vaccine was being administered. The researchers at the Kirsehir Training and Research Hospital in Turkey will apply their findings to healthy newborns who are placed adjacent to their moms in the postpartum ward. The researchers have experience in neonatal critical care nursing and are qualified in therapeutic touch.

DETAILED DESCRIPTION:
After birth, the fetus undergoes a process of transformation from its diverse physiological and anatomical state during the intrauterine period. During the first 28 days of life, every newborn's bodily systems and functions continue to evolve in an effort to adjust to the extrauterine world.

With the right treatment, extrauterine adaption can be ensured for the newborn during this dangerous time. Many invasive procedures for diagnosis and prevention are part of healthy newborn care, and they are crucial for maintaining health once early extrauterine adaption is achieved. These invasive procedures include blood sugar testing, intramuscular injections, heel blood collection, and blood collection from peripheral veins.

Contrary to popular assumption, neonates have more sensitive pain perception, and it is well recognized that discomfort in newborns can lead to a variety of issues. The American Academy of Pediatrics states that pain is an unpleasant emotional and sensory experience brought on by actual or anticipated texture.

Infants experience pain to the same extent as adults do. So much so that pain in babies has been linked to a wide range of both immediate and long-term consequences, including altered physiological parameters, issues with nutrition and sleep, chronic pain syndrome, difficulty focusing, anxiety, cognitive behavioral disorders, adjustment disorder, and growth retardation. Each and every newborn is entitled to pain relief and reduction.

Avoiding painful interventions is the most crucial tactic in the management of newborn pain. It is impossible to avoid the necessity for therapeutic and diagnostic procedures, though. As such, pain reduction and elimination are crucial. According to studies, non-pharmacological techniques used on infants undergoing invasive operations are successful in reducing discomfort, pain, and restlessness while enhancing comfort. Numerous non-invasive, non-pharmacological techniques are employed for this goal. Among the non-invasive, non-pharmacological techniques include breastfeeding, nursing, therapeutic touch, skin-to-skin contact, wrapping, swaddling, music therapy, and white noise.

The Hepatitis-B vaccine is among the first invasive therapies administered to infants. Research indicates that pain scores are positively impacted by canopy touch. Skin-to-skin contact is achieved by a number of techniques. The most popular is kangaroo care, which is given to mothers nude on their chests.Gentle human touch is another technique used to lessen pain during invasive operations (GHT). GHT is a soothing tactile stimulation that doesn't involve touching or rubbing. Numerous research have examined GHT's impact and discovered that it effectively reduces pain.

In order to ensure patients' comfort and minimize the harmful effects of uncomfortable treatments, nurses play a crucial role. supplemental medical attention Basic nursing procedures have built-in techniques that help lessen the discomfort of intrusive interventions. Thus, the purpose of this study was to compare the effects of the two applications and assess the impact of kangaroo care and GHT on pain, duration of crying, and physiological parameters during the administration of the Hepatitis-B vaccine to neonates.Research Design: This study was designed as a randomized controlled experimental design to assess the impact of GHT and kangaroo care on newborn infants' pain, length of crying, and physiological parameters during the administration of the Hepatitis-B vaccine. Location and Study Features: The Gynecology and Obstetrics Service of the Kırşehir Training and Research Hospital in Turkey will be the site of this research. The ward has twelve nurses and twenty-eight beds. Every year, on average, 1000 people are born. The universe and study sample: To decide how many newborns should be in the research sample, a power analysis will be done at the start of the study. Upon reviewing the pertinent literature, it becomes evident that comparable research have utilized samples.Analyzing the pertinent literature reveals that research with similar designs have sampled between 30-35 groups. Research will be assessed in relation to the comparable research sample. The G*power tool will then be used by a statistician to do a power analysis. Study Universe and Sample: The number of newborn newborns to be included in the research sample will be determined at the outset of the study through a power analysis. Analyzing the pertinent literature reveals that research with similar designs have sampled between 30-35 groups. Research will be assessed in relation to the comparable research sample. The G*power tool will then be used by a statistician to do a power analysis.

At least thirty babies will be included in each of the three groups that will be randomly assigned, along with a control group. The sample group will be randomly assigned numbers ranging from 1 to 90 using the web software www.randomizer.org to identify the groups to which the newborns will be placed.A statistician will conduct post-power analysis once there are ninety samples.

Data collecting Form is the first data collecting tool. 1. The researcher scanned the literature to generate this form. It asks about the parents' sociodemographic details as well as the newborn's birth weight, height, head circumference, first and fifth Apgar scores, gestational week, and gender.

2. The NIPS (Neonatal Infant Pain Scale) 3. Registration Form for Application This form is used to record the groups' physiological parameters and NIPS score before, during, and after the hepatitis-B vaccination procedure.

Methods and Approach to Be Used Mothers who are calm before giving birth will be invited to participate in the study. Mothers who volunteer to participate in the research and meet the eligibility requirements will have their written consent obtained.

Both the mother and the child are expected to be stable following delivery. Prior to the surgery, the newborns' physiological parameters (heart rate and SpO2) will be monitored by attaching a neonatal probe to the pulse oximetry.

Next, the groups selected by randomization will receive GHT with Gentle Human Touch (Group 1), Kangaroo Care (Group 2), and Control Group (Group 3). Without affecting the control group, the researcher will conduct the GHT and provide kangaroo care with the moms of the infants. The same nurse will give each baby the hepatitis-B vaccination. A neonatal nurse will use a stopwatch to monitor the newborn's screaming times during the process.

ELIGIBILITY:
Inclusion Criteria:

Gestational week between 38-42,

* Born at 38 weeks or above and with a body weight of >2500 grams,
* Apgar score 1st and 5th 7 and above per minute,
* Mothers who speak and speak Turkish

Exclusion Criteria:

* Congenital anomaly
* Hospitalization of the baby in the neonatal intensive care unit after birth
* Mothers with hepatitis B vaccine refusal
* Mothers who do not have kangaroo care

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
pain level | before vaccination/ immediately after vaccination
  The newborn's pain assessment will be measured by NIPS. In the scale, the baby's facial expression (0-1 point), crying (0-2 points), breathing pattern (0-1 point), arm movements (0-1 point), leg movements (0-1 point) and alertness ( Scores between 0-7 are given according to 0-1 points). An increase in the score on the scale indicates a higher severity of pain.

SECONDARY OUTCOMES:
newborn crying duration | immediately after vaccination
  The newborn's crying duration will be measured and recorded with a stopwatch
Saturation | before vaccination/ immediately after vaccination
  A portable pulse oximeter device will be used. saturation will be recorded and evaluated.
Heart rate | before vaccination/ immediately after vaccination
  A portable pulse oximeter device will be used.
Respiratory rate | before vaccination/ immediately after vaccination
  A portable pulse oximeter device will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uematsu H, Sobue I. Effect of music (Brahms lullaby) and non-nutritive sucking on heel lance in preterm infants: A randomized controlled crossover trial. Paediatr Child Health. 2019 Feb;24(1):e33-e39. doi: 10.1093/pch/pxy072. Epub 2018 Jul 24. PMID 30792607
- [Background] Im H, Kim E. Effect of Yakson and Gentle Human Touch versus usual care on urine stress hormones and behaviors in preterm infants: a quasi-experimental study. Int J Nurs Stud. 2009 Apr;46(4):450-8. doi: 10.1016/j.ijnurstu.2008.01.009. Epub 2008 Mar 18. PMID 18353332
- [Background] Dur S, Caglar S, Yildiz NU, Dogan P, Guney Varal I. The effect of Yakson and Gentle Human Touch methods on pain and physiological parameters in preterm infants during heel lancing. Intensive Crit Care Nurs. 2020 Dec;61:102886. doi: 10.1016/j.iccn.2020.102886. Epub 2020 Jun 27. PMID 32601011
- [Background] Huang Q, Lai X, Liao J, Tan Y. Effect of non-pharmacological interventions on sleep in preterm infants in the neonatal intensive care unit: A protocol for systematic review and network meta-analysis. Medicine (Baltimore). 2021 Oct 29;100(43):e27587. doi: 10.1097/MD.0000000000027587. PMID 34713833
- [Background] Sezer Efe Y, Erdem E, Caner N, Gunes T. The effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing. Complement Ther Clin Pract. 2022 Aug;48:101622. doi: 10.1016/j.ctcp.2022.101622. Epub 2022 Jun 22. PMID 35759976